CLINICAL TRIAL: NCT03448497
Title: Retrospective Chart Review Study of First-line Treatment Patterns and Clinical Outcomes in Patients With Advanced (Unresectable or Metastatic) Melanoma in the United Kingdom
Brief Title: Study of First-line Treatment Patterns and Clinical Outcomes in Patients With Advanced Melanoma in the United Kingdom
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9TW
Record Dates: First submitted 2018-02-12; First posted 2018-02-28 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Advanced Melanoma patients who intiated first-line therapy: patients who initiated any first-line therapy for advanced melanoma and had not previously received treatment for their advanced disease
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
The purpose of this study is to describe the first-line therapy landscape for patients with advanced melanoma and to describe clinical outcomes and healthcare resource utilization in a subset of treatment-naïve patients who initiated nivolumab + ipilimumab combination therapy.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patient has medical chart documentation of advanced (unresectable or metastatic) melanoma.
* Patient initiated a first-line therapy for the treatment of advanced melanoma during the eligibility period (01 July 2016 to 01 July 2017; index event).
* Patient did not receive systemic treatment for their advanced (unresectable or metastatic) melanoma prior to index event
* Patient initiated first-line therapy at least six months before the date their chart abstraction initiated

Exclusion Criteria:

* Patient was enrolled in an investigational drug clinical trial or participating in medical research judged to directly affect how the patient was being monitored/treated while receiving first-line therapy
* Patient had another active concurrent malignancy other than advanced melanoma, which required systemic treatment at the time of index event
* Part or all of the patient's first-line treatment was received at a different site and the patient's medical chart pertaining to this care is not accessible
* Patient medical chart is missing, empty, or not retrievable

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes treatment-naïve patients with advanced (unresectable or metastatic) melanoma who initiated first-line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Best Overall Response (BOR) rate | Up to 18 months
  In a subset of patients treated with first-line nivolumab + ipilimumab combination therapy

SECONDARY OUTCOMES:
Distribution of patient demographic characteristics | At baseline
  Including age, sex, ethnic group, height, weight, and BMI
Prior melanoma treatment history | At baseline
  Type of intervention used to treat melanoma
Serum concentration of lactate dehydrogenase (LDH) | At baseline
Eastern Cooperative Oncology Group (ECOG) score | Up to 18 months
Distribution of first-line treatment patterns | Up to 18 months
  Details on Treatment Patterns will be summarized using descriptive statistics
Distribution of subsequent therapy line treatment patterns | Up to 18 months
  Details on Treatment Patterns will be summarized using descriptive statistics
Progression Free Survival (PFS) | Up to 18 months
  Time from first-line initiation until disease progression or death in a subset of patients treated with first-line nivolumab + ipilimumab combination therapy
Treatment-Free Interval (TFI) | Up to 18 months
  Time from nivolumab + ipilimumab combination therapy discontinuation to date of progressive disease in a subset of patients treated with first-line nivolumab + ipilimumab combination therapy
Overall Survival (OS) | Up to 18 months
  Time from treatment initiation until death in a subset of patients treated with first-line nivolumab + ipilimumab combination therapy
Distribution of PD-L1 threshold | At baseline
  PD-L1 threshold used for first-line treatment selection in patients where PD-L1 was tested
Incidence of adverse events of Special interest(AESI) | Up to 18 months
  in a subset of patients receiving nivolumab + ipilimumab combo therapy. AESIs include select gastrointestinal, renal, pulmonary, hepatic, endocrine, skin, neurological, and infusion reaction.
Incidence of serious adverse events (SAE) | Up to 18 months
  in a subset of patients receiving nivolumab + ipilimumab combo therapy. SAE defined as Common Terminology Criteria for Adverse Events (CTCAE) grades 3+ adverse events
Distribution of AESI management | up to 18 months
  In a subset of patients receiving Nivo + Ipi combo therapy
melanoma related healthcare resource utilization (HCRU) | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm